CLINICAL TRIAL: NCT03508726
Title: Phase 1b/2 Neoadjuvant High Dose Ascorbate With Concurrent Preoperative Radiation in Patients With Locally Advanced Soft Tissue Sarcomas of Extremity, Trunk and Retroperitoneum
Brief Title: High Dose Ascorbate With Preoperative Radiation in Patients With Locally Advanced Soft Tissue Sarcomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mohammed Milhem (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Mohammed Milhem, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201901810
Record Dates: First submitted 2018-04-13; First posted 2018-04-26 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Soft Tissue Sarcoma
Keywords: Sarcoma; Soft tissue
MeSH Terms: conditions — Sarcoma | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I dose escalation cohort (Experimental): Participants will receive radiation therapy over 5 weeks, during which time they will be receiving ascorbate infusions three times a week. Ascorbate infusions will be continued until the end of radiation therapy. Surgery will be performed 4-6 weeks from the end of radiation.
  Interventions: Drug: Ascorbate
- Phase II Cohort (Experimental): Participants will receive radiation therapy over 5 weeks, during which time they will be receiving intravenous (IV) ascorbate infusions three times a week. Ascorbate infusions will be continued until the end of radiation therapy. Surgery will be performed 4-6 weeks from the end of radiation.
  Interventions: Drug: Ascorbate

INTERVENTIONS:
Drug: Ascorbate — Phase 1 dose escalation:
  75gm IV three times a week
  Phase II portion:
  75gm IV three times a week if no dose limiting toxicities are experienced in the Phase I portion. Otherwise, ascorbate dose will be deescalated to 62.5 gm IV
  Other Names: Ascorbic Acid; Vitamin C; Pharmacological ascorbate

SUMMARY:
This is a single-arm open-label phase Ib/II clinical study assessing the efficacy of concurrent high dose ascorbate in combination with radiotherapy in patients with locally advanced, resectable, high grade sarcomas.

DETAILED DESCRIPTION:
Phase Ib:

The phase Ib portion of this study is to ensure the safety and tolerability of high dose ascorbate in combination with external beam radiation therapy (EBRT) as assessed by incidence of dose-limiting toxicities (DLT). EBRT will be given at the standard dose for resectable soft tissue sarcomas according to the NCCN sarcoma guidelines.2 Patients will receive 50 Gy over 5 weeks, during which time they will be receiving three times a week IV high dose ascorbate. IV ascorbate infusions will be continued until the end of radiation therapy. Surgery will be performed 4-6 weeks from the end of radiation to allow for adequate tissue healing and resolution of acute toxicities.

Phase 2:

The phase 2 part of the study will provide an estimate of the relative treatment effect of pharmacological ascorbate in combination with preoperative EBRT in subjects with locally advanced, resectable, extremity, trunk or retroperitoneal high grade sarcomas, as measured by pathological response rates.

As above, patients will receive the first dose of pharmacological ascorbate intravenously on day 1 of week 1 provided no reactions are seen to the test dose. This will be followed by 3 times a week dosing at Dose 0 until completion of EBRT. Standard doses of radiation for resectable soft tissue sarcomas according to the NCCN sarcoma guidelines will be administered.2 Patients will receive preoperative radiation at a dose of 50 Gy over 5 weeks starting on week 1 day 1. Subjects will be followed either by clinic visit or phone contact every 12 weeks for approximately 24 months after the end of the treatment phase, at which time the initial survival data and disease recurrence will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or subject's legally acceptable representative has provided informed consent.
2. Histologically confirmed diagnosis of locally advanced soft tissue sarcoma of extremity, trunk or retroperitoneum that is unresectable with clear wide margins, for which preoperative radiotherapy is considered appropriate

   - Including metastatic (stage IV) disease for which radiotherapy and surgical resection of the primary tumor are indicated.
3. Patients with locally recurrent sarcoma after surgery alone are eligible for enrollment if other inclusion criteria are met.
4. Patients do not have histologic subtypes: GIST, Desmoid, Ewing sarcoma, bone sarcomas and Kaposi sarcoma.
5. Age ≥18 years.
6. Patients with a history of non-melanomatous skin cancer, in situ carcinoma, or low-risk prostate cancer can be enrolled.
7. ECOG performance status </=1.
8. Tolerate one test dose (15g) of ascorbate.
9. Patient must have measurable disease:

   * Tumor size at least >/= 5 cm in the longest diameter as measured by CT scan or MRI for which radiation is feasible and indicated.

Exclusion Criteria:

1. Inadequate organ function within 21 days of Day 1 of study as defined by:

   * Hemoglobin < 9.0 g/dL
   * Absolute neutrophil count (ANC) </= 1500 per mm3
   * Platelet count </= 100,000 per mm3
   * Total bilirubin >/= 1.5 × ULN. Subjects with direct bilirubin < ULN with total bilirubin levels > 1.5 X ULN will not be excluded.
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × ULN
   * Alkaline phosphatase > 2.5 × ULN
   * PT (or INR) and PTT (or aPTT) >/= 1.5 × ULN
   * Creatinine > 2.0 × ULN
2. G6PD (glucose-6-phosphate dehydrogenase) deficiency.
3. Prior history of symptomatic oxalate kidney stones within the last year.
4. Prior radiation therapy in excess of 20 Gy to the site of the current diagnosis of sarcoma. No overlap with prior radiation fields in excess of 20 Gy is allowed.
5. Prior history of receiving pharmacological ascorbate.
6. Patients actively receiving insulin therapy and needing daily fingerstick for glucose monitoring.
7. Concurrent, clinically significant, active malignancies within two years of study enrollment.
8. Female subjects who are pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of study treatment.
9. Female subjects of childbearing potential or male subjects who are unwilling to use 2 highly effective methods of contraception during study treatment and through 3 months after the last dose of study treatment.
10. Currently receiving treatment in another invasive investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s).
11. Patients who are on the following drugs and cannot have a drug substitution: flecainide, methadone, amphetamines, quinidine, and chlorpropamide. High dose ascorbic acid may affect urine acidification and, as a result, may affect clearance rates of these drugs.
12. Known CNS disease, except for treated brain metastasis: Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
13. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ascorbate.
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Known HIV-positive and hepatitis B & C individuals. High-dose ascorbate acid is a known CYP450 3A4 inducer, which results in lower serum levels of antiretroviral drugs.
16. Patients who are on warfarin and cannot have a drug substitution or who decline the drug substitution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2024-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MBBS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Principal Investigator's and Sub-Investigator's clinics at Holden Comprehensive Cancer Center.
Groups:
- Phase I: Ascorbate 75 mg IV Infusion: Participants will receive radiation therapy over 5 weeks, during which time they will be receiving ascorbate infusions three times a week. Ascorbate infusions will be continued until the end of radiation therapy. Surgery will be performed 4-6 weeks from the end of radiation.
- Phase II: Ascorbate 75 mg IV Infusion: Participants will receive radiation therapy over 5 weeks, during which time they will be receiving intravenous (IV) ascorbate infusions three times a week. Ascorbate infusions will be continued until the end of radiation therapy. Surgery will be performed 4-6 weeks from the end of radiation.
Period: Overall Study
Arm/Group | Phase I: Ascorbate 75 mg IV Infusion | Phase II: Ascorbate 75 mg IV Infusion
Started | 6 | 19
Completed | 6 | 18
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Ascorbate 75 mg IV Infusion: Participants will receive radiation therapy over 5 weeks, during which time they will be receiving ascorbate infusions three times a week. Ascorbate infusions will be continued until the end of radiation therapy. Surgery will be performed 4-6 weeks from the end of radiation.
  All participants received 75 mg Ascorbate IV dose three times a week.
- Phase II: Ascorbate 75 mg IV Infusion: Participants will receive radiation therapy over 5 weeks, during which time they will be receiving intravenous (IV) ascorbate infusions three times a week. Ascorbate infusions will be continued until the end of radiation therapy. Surgery will be performed 4-6 weeks from the end of radiation.
  All participants received 75 mg Ascorbate IV dose three times a week.
- Total: Total of all reporting groups
Arm/Group | Phase I: Ascorbate 75 mg IV Infusion | Phase II: Ascorbate 75 mg IV Infusion | Total
Number analyzed (Participants) | 6 | 19 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 2 | 14 | 16
Age, Continuous [Mean (Full Range); unit: years] | 60 [39 to 85] | 67 [42 to 87] | 65 [39 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 2 | 12 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 19 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 19 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 19 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced Dose Limiting Toxicities (DLTs) Using CTCAE, Version 4.0
Description: To examine the toxicity related to the therapy by measuring the number attributed adverse event (definite, probable or possible) according to CTCAE version 4.0.
Time Frame: Start of treatment up to 4 weeks after the last ascorbate infusion
Population: 6 participants enrolled in the Phase 1 dose escalation portion of the trial and were assessed for dose limiting toxicities. All participants received 75 mg Ascorbate IV dose three times a week.
Measure: Number; unit: participants
Groups:
- Phase I: Ascorbate 75 mg IV Infusion: Patients will receive radiation therapy over 5 weeks, during which time they will be receiving ascorbate infusions three times a week. Ascorbate infusions will be continued until the end of radiation therapy. Surgery will be performed 4-6 weeks from the end of radiation.
Arm/Group | Phase I: Ascorbate 75 mg IV Infusion
Number analyzed (Participants) | 6
participants | 0

2. Primary Outcome: Number of Participants With Pathologic Tumor Necrosis ≥ 95% Following Concurrent Radiation Therapy and Ascorbate
Description: To estimate the efficacy of neoadjuvant ascorbate and radiotherapy as assessed by the pathological complete response rates (pCR) in subjects with locally advanced high grade soft tissue sarcomas.
Time Frame: Start of treatment up to 6 weeks after the last ascorbate infusion
Population: 6 participants enrolled to the Phase I portion and were assessed for pCR. 18 participants were enrolled to the Phase II portion and assessed by for pCR via pathological reading. All participants in both Phase cohorts received 75 mg Ascorbate IV dose three times a week.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ascorbate 75 mg IV Infusion | Phase II: Ascorbate 75 mg IV Infusion
Number analyzed (Participants) | 6 | 18
Participants | 2 | 1

3. Secondary Outcome: Disease Progression as Measured by Time to Disease Progression (TTP)
Description: Time to disease progression (TTP) is defined as the time from enrollment until objective tumor progression including local and distant recurrences.
Time Frame: Enrollment or start of treatment up to 2 years following end of treatment
Reporting Status: Not Posted

4. Secondary Outcome: Overall Response Rate as Measured by RECIST 1.1
Description: Overall response rate (ORR) preoperative as measured by RECIST 1.1 or a later tool for monitoring disease progression.
Time Frame: Enrollment or start of treatment up to 2 years following end of treatment
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival Estimated Using the Kaplan-Meier Method
Description: Overall survival (OS) rate data gathered through passive chart review, phone call or scheduled follow-up visit and estimated using the Kaplan-Meier Method.
Time Frame: Enrollment or start of treatment up to 2 years following end of treatment
Reporting Status: Not Posted

6. Secondary Outcome: Skin Toxicity
Description: Pathologist to grade radiation related skin toxicity overlying the tumor as compared to historical controls. Binomial exact tests will be utilized to identify differences in wound complication and Grade 3-4 dermatitis rates compared to historical controls.
Time Frame: Within two years following end of treatment
Reporting Status: Not Posted

7. Secondary Outcome: Labile Iron
Description: To measure labile iron using T2* imaging sequence on MRI pre and post ascorbate treatments and compare with serum iron measurements
Time Frame: Within two years following end of treatment
Reporting Status: Not Posted

8. Secondary Outcome: Evaluate Diffusion Weighted Imaging Sequences
Description: To evaluate diffusion weighted imaging sequences on MRI in pre and post treatment tumors and correlate it with necrosis and survival
Time Frame: Within two years following end of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For any experience or condition that meets the definition of a adverse event (AE), recording of the event must begin after signing of Informed Consent Form and continue through the 30-day follow up period after treatment is discontinued, up to 12 weeks.
Arm/Group | Phase I: Ascorbate 75 mg IV Infusion | Phase II: Ascorbate 75 mg IV Infusion
All-Cause Mortality (participants affected / at risk) | 0/6 | 5/19
Serious Adverse Events (participants affected / at risk) | 0/6 | 4/19
Other Adverse Events (participants affected / at risk) | 6/6 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Ascorbate 75 mg IV Infusion (N=6) | Phase II: Ascorbate 75 mg IV Infusion (N=19)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Ascorbate 75 mg IV Infusion (N=6) | Phase II: Ascorbate 75 mg IV Infusion (N=19)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 7 (10)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (6) | 9 (11)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 5 (6)
Fatigue (General disorders) | 3 (3) | 5 (5)
Fever (General disorders) | 0 (0) | 2 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 3 (5)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (3) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Alanine aminotransferase increased (Investigations) | 2 (3) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (6)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 3 (4) | 8 (26)
Lymphocyte count decreased (Investigations) | 4 (4) | 7 (14)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 3 (3)
Weight loss (Investigations) | 0 (0) | 2 (4)
White blood cell decreased (Investigations) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 6 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 5 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 6 (9)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (8) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT03508726/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT03508726/ICF_001.pdf